CLINICAL TRIAL: NCT01292655
Title: Phase 1 Ascending Multiple-Dose Study to Evaluate the Safety, Pharmacokinetics (PK) and Pharmacodynamics (PD) of BMS-906024 in Subjects With Advanced Solid Tumors
Brief Title: Study to Evaluate the Safety and Tolerability of IV Doses of BMS-906024 in Subjects With Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA216-001
Record Dates: First submitted 2011-01-26; First posted 2011-02-09 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — BMS-906024

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A1 (Escalation): BMS-906024 (Experimental): BMS-906024 solution intravenously as specified
  Interventions: Drug: BMS-906024
- Arm A2 (Expansion): BMS-906024 (Experimental): BMS-906024 solution intravenously as specified
  Interventions: Drug: BMS-906024
- Arm B1 (Escalation): BMS-906024 (Experimental): BMS-906024 solution intravenously as specified
  Interventions: Drug: BMS-906024
- Arm B2 (Expansion): BMS-906024 (Experimental): BMS-906024 solution intravenously as specified
  Interventions: Drug: BMS-906024

INTERVENTIONS:
Drug: BMS-906024
  Other Names: BMS-906024 (Notch inhibitor)

SUMMARY:
The purpose of this study is to identify a safe and tolerable dose of BMS-906024 in subjects with advanced or metastatic solid tumors who no longer respond to or have relapsed from standard therapies.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Subjects with advanced or metastatic solid tumors (non-hematologic refractory to or relapsed from standard therapies or for which there is no known effective treatment during dose escalation
* Subjects with squamous non-small cell lung cancer and triple-negative breast cancer or other solid tumor types for which Notch activation has been demonstrated (such as pancreatic, ovarian and melanoma) during dose expansion
* Biopsy accessible tumor (may be waived under certain circumstances)
* Life expectancy of at least 3 months
* Eastern Cooperative Oncology Group (ECOG) 0-1
* Adequate organ and bone marrow function

Exclusion Criteria:

* Infection
* Elevated triglycerides
* Gastrointestinal (GI) disease with increased risk of diarrhea [e.g. inflammatory bowel disease (IBD)]
* Taking medications known to increase risk of Torsades De Pointes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2011-03-03 (Actual); Primary Completion 2017-06-22 (Actual); Study Completion 2017-06-22 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events as a measure of safety and tolerability | Weekly assessments until study discontinuation due to disease progression or unacceptable adverse event as well as an assessment 30 day after treatment discontinuation with an average time on study expected to be <1 year

SECONDARY OUTCOMES:
Tumor assessments using response evaluation criteria in solid tumors (RECIST) v1.1 | Tumor assessments at least every 8 weeks during treatment period
PD changes from baseline in the expression of Notch pathway-related genes in surrogate tissues (peripheral blood cells) and tumor biopsies | PD changes from baseline during the first 4-5 weeks of dosing
PK parameters for BMS-906024 and its metabolite BMS-911557, maximum observed concentration (Cmax) | PK at multiple time points during the first 8 weeks of dosing
PK parameters for BMS-906024 and its metabolite BMS-911557, minimum observed concentration (Cmin) | PK at multiple time points during the first 8 weeks of dosing
PK parameters for BMS-906024 and its metabolite BMS-911557, time to reach maximum observed concentration (Tmax) | PK at multiple time points during the first 8 weeks of dosing
PK parameters for BMS-906024 and its metabolite BMS-911557, terminal phase elimination half-life (T-Half) | PK at multiple time points during the first 8 weeks of dosing
PK parameters for BMS-906024 and its metabolite BMS-911557, accumulation index (AI) | PK at multiple time points during the first 8 weeks of dosing
PK parameters for BMS-906024 and its metabolite BMS-911557, area under the concentration-time curve (AUC) | PK at multiple time points during the first 8 weeks of dosing

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (8):
- United States (6):
  - Anthony El-Khoueiry, Md, Los Angeles, California
  - Winship Cancer Institute., Atlanta, Georgia
  - Wayne State University, Detroit, Michigan
  - University Of Mississippi Medical Center, Jackson, Mississippi
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - The Methodist Hospital Research Institute, Houston, Texas
- Local Institution, Parkville, Victoria, Australia
- Local Institution, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Chan D, Kaplan J, Gordon G, Desai J. Activity of the Gamma Secretase Inhibitor AL101 in Desmoid Tumors: A Case Report of 2 Adult Cases. Curr Oncol. 2021 Sep 21;28(5):3659-3667. doi: 10.3390/curroncol28050312. PMID 34590610
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx